CLINICAL TRIAL: NCT00261781
Title: Does Home-based Treadmill Training Improve Walking Capacity and Quality of Life in People With Early to Mid-stage Parkinson's Disease?
Brief Title: Walking Capacity in Parkinson's Disease (PD-Walk)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 20 subjects completed for a pilot, further funding required to continue study
Sponsor: Natalie Allen (Other)
Collaborators: South West Sydney Local Health District (Other)
Responsible Party: Sponsor-Investigator, Natalie Allen, Dr Natalie allen, University of Sydney
Organization: University of Sydney (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U3189
Record Dates: First submitted 2005-12-01; First posted 2005-12-05 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2015-05

CONDITIONS: Idiopathic Parkinson's Disease
Keywords: Treadmill; Walking; Exercise; Automaticity; Quality of Life
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treadmill training (Experimental): Home-based treadmill training
  Interventions: Behavioral: Treadmill training
- Usual care (No Intervention): Control group

INTERVENTIONS:
Behavioral: Treadmill training — Walking on a treadmill 3 times per week for 6 weeks
  Arms: Treadmill training

SUMMARY:
The major aim of this study is to determine the efficacy of a home-based treadmill walking program in improving walking capacity and quality of life in people with early mid-stage Parkinson's disease(PD).

DETAILED DESCRIPTION:
After Alzheimer's disease, Parkinson's disease (PD) is the most common degenerative neurological condition suffered by Australians, with more than 30,000 Australians having PD at any one time (Parkinson's Australia). Hypokinesia, ie, reduced speed and amplitude of movement, is a major impairment of motor control affecting walking in people with PD. Over time, the development of slow, shuffling walking contributes to loss of independence and falls, with devastating consequences for individuals with PD and their families(Ashburn et al, 2001, Playfer 2001). Any decrease or delay in disability will reduce the personal and financial costs to individuals with PD, their families, health care resources and the community.

A number of previous studies suggest exercise capacity and exercise habits are positively correlated. In people with mild Parkinson's disease (Canning et al 2005), walking capacity, measured as distance walked in the 6-min walk test, correlated with the amount of walking (r=.64, p<0.01) performed each week. Similarly, in an earlier study of people with mild to moderate Parkinson's disease, regular exercise was associated with better exercise capacity (Canning et al 1997). It appears, therefore, that proactive intervention aimed at developing good exercise habits in sedentary individuals with early to mid-stage Parkinson's disease has the potential to reduce or delay walking difficulties.

This study aims to establish the efficacy of a home-based treadmill walking program in providing an early intervention which addresses the primary motor control impairment of hypokinesia, while at the same time maintaining or improving exercise capacity.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of idiopathic Parkinson's disease
* aged 30-80 years old
* subjective disturbance of gait and / or Unified Parkinson's disease rating scale (UPDRS) gait subscore of 1
* sedentary, defined as performing less than 2 hours / week of leisure-time physical activity over the prior 3 months
* have adapted to their current anti-Parkinsonian medication for at least 2 weeks

Exclusion Criteria:

* motor fluctuations or dyskinesias which are disabling
* require the use of a walking aid
* more than one fall in the last 12 months
* Mini-Mental State Examination score of <24
* exhibit other neurological or musculoskeletal conditions affecting walking
* chest pain at rest or during exercise in the last 3 months, or heart attack, angioplasty or heart surgery in the last 6 months

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-05; Primary Completion 2006-12 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Distance walked in 6 minutes | study entry (0 weeks), 7 and 13 weeks

SECONDARY OUTCOMES:
Unified Parkinson's disease Rating Scale (UPDRS) - motor examination | 0, 7 and 13 weeks
The Parkinson's disease Questionnaire (PDQ-39 | 0, 7 and 13 weeks
Walking Automaticity, determined as the velocity of walking 10m while performing a concurrent (cognitive or cognitive + physical) task expressed as a percentage of the velocity of walking 10m without performing the concurrent task. | 0, 7 and 13 weeks
Walking consistency determined as the co-efficients of variation for stride time and stride length recorded during the 6 minute walk test. | 0, 7 and 13 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Colleen G Canning, PhD, Principal Investigator — University of Sydney
Locations (1):
- Westmead Hospital, Sydney, New South Wales, Australia

REFERENCES:
- [Background] Ashburn A, Stack E, Pickering RM, Ward CD. A community-dwelling sample of people with Parkinson's disease: characteristics of fallers and non-fallers. Age Ageing. 2001 Jan;30(1):47-52. doi: 10.1093/ageing/30.1.47. PMID 11322672
- [Background] Canning CG, Alison JA, Allen NE, Groeller H. Parkinson's disease: an investigation of exercise capacity, respiratory function, and gait. Arch Phys Med Rehabil. 1997 Feb;78(2):199-207. doi: 10.1016/s0003-9993(97)90264-1. PMID 9041903
- [Background] Playfer JR. Falls and Parkinson's disease. Age Ageing. 2001 Jan;30(1):3-4. doi: 10.1093/ageing/30.1.3. No abstract available. PMID 11322669
- [Result] Canning CG, Allen NE, Dean CM, Goh L, Fung VS. Home-based treadmill training for individuals with Parkinson's disease: a randomized controlled pilot trial. Clin Rehabil. 2012 Sep;26(9):817-26. doi: 10.1177/0269215511432652. Epub 2012 Jan 18. PMID 22257506